CLINICAL TRIAL: NCT02566421
Title: Precision Medicine for Patients With Malignancy at the Comprehensive Cancer Center of Wake Forest University
Brief Title: Genomic Sequencing in Determining Treatment in Patients With Metastatic Cancer or Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Assessing Feasibility
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00033598; NCI-2015-01373 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01615; IRB00033598; CCCWFU # 01615 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-09-14; First posted 2015-10-02 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Metastatic Neoplasm; Recurrent Neoplasm; Recurrent Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer; Unresectable Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (precision medicine) (Experimental): Patients receive treatment based on the results of their genomic sequencing analyses.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Targeted Therapy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Targeted Therapy — Receive treatment based on genomic sequencing

SUMMARY:
This pilot clinical trial studies patients' genomic sequencing in determining specific treatments, also called Precision Medicine, in patients with cancer that has spread to other parts of the body (metastatic) and/or cannot be removed by surgery. Examining the genetic code of a patient's tumor, a mutation (a change in the deoxyribonucleic acid [DNA] sequence of a cell or gene) may be identified and matched with available treatment that targets the mutated gene or an alternative treatment that may provide benefit for the patient with the mutation identified. Precision medicine may impacts patient's response to treatment by targeting specific mutations and may increase survival and improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of implementing a Precision Oncology protocol in the treatment of patients who undergo genomic sequencing.

SECONDARY OBJECTIVES:

I. To determine treatment response rates in patients who receive targeted treatment versus those who do not receive targeted treatment.

II. To assess survival in patients who receive targeted treatment versus those who do not receive targeted treatment.

III. To assess changes in patient-reported outcomes in patients who receive targeted treatment versus those who do not receive targeted treatment.

IV. To perform exploratory statistical genetic and bioinformatics analyses using the data derived from the genomic sequencing to catalogue additional important variants and determine whether there are any patterns or associations among patient level risk factors, their outcomes and genomic information that was not identified by the original genomic sequencing analyses.

OUTLINE:

Patients receive treatment based on the results of their genomic sequencing analyses.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable cancer for which there are genomic drivers with corresponding Food and Drug Administration (FDA) approved or experimental drugs available, e.g. non-small cell lung cancer; and/or patients with histologically confirmed metastatic malignancy that have failed standard treatment or cannot tolerate standard treatment as deemed by the treating physician
* Malignancy must be measureable as per appropriate guidelines
* Patients who are willing to provide a specimen for genomic sequencing

  * Preferred method:

    * Tumor cell sample available and of sufficient quantity in the Tumor Tissue Shared Resource or patients who are willing to undergo additional tissue collection for tumor genomic sequencing through FoundationOne; available specimens must have been harvested within two years to be eligible
  * Alternative method:

    * Patients who are unwilling or unable to provide a tumor tissue sample and who undergoes Guardant360 sequencing may be considered eligible by the treating physician
  * Patients who have already had their specimens sent for genomic sequencing are eligible provided they have not received their sequencing results at the time of enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absence of clinically relevant liver or kidney failure as deemed by the treating physician
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diminished mental capacity or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Feasibility in terms of the ability to monitoring patient outcomes across separate treatment protocols and study teams. | Up to 2 years
  Typical patient outcome measures will necessarily vary by disease, so survival will be the overarching outcome measure.
Proportion of patients enrolled on this protocol who are subsequently enrolled in a clinical trial based on the results of the genomic sequencing | Baseline
Proportion of patients enrolled on this protocol who have a clinical trial identified for them to be enrolled in based on the results of the genomic sequencing | Baseline
  The observed proportion and corresponding 95% confidence intervals will be estimated.
Proportion of patients with an actionable mutation | Baseline
  Each patient enrolled will be dichotomized into either having a clinical trial identified (yes/no) that the results of their genomic sequencing suggests. The observed proportion and corresponding 95% confidence intervals will be estimated.
Feasibility in terms of the ability to monitoring patient adverse events across separate treatment protocols and study teams. | Up to 2 years

SECONDARY OUTCOMES:
Change in patient-reported symptoms of cancer and cancer treatment, as assessed by the MD Anderson Symptom Inventory | Baseline to up to 48 weeks
Patient's perceived quality care, as assessed by 3 items adapted from Arora, et al | Up to up to 48 weeks
Patient's satisfaction with treatment decision-making and decisional regret, as assessed by an adapted Satisfaction with Decision scale | Up to up to 48 weeks
Self-perceived burden, as assessed by the Self-Perceived Burden Scale-Short form for measuring chronic disease patients' feelings of being a burden on their caregivers | Up to up to 48 weeks
Survival rate in patients who receive targeted treatment versus those who do not receive targeted treatment | Up to 6 months
  Kaplan Meier curves will be estimated and groups will be compared using Log-Rank tests. These analyses will be performed across all disease sites and then stratified by disease site.
Survival rate in patients who receive targeted treatment versus those who do not receive targeted treatment | Up to 12 months
  Kaplan Meier curves will be estimated and groups will be compared using Log-Rank tests. These analyses will be performed across all disease sites and then stratified by disease site.
Treatment response rates in patients who receive targeted treatment versus those who do not receive targeted treatment | Up to 2 years
  For each patient a clinical response assessment will be ascertained and compared between groups. 95% confidence intervals will be estimated for the response rates (with stable disease [SD], partial response [PR] and complete response [CR] pooled together) and the repeated with PR and CR pooled together.

OTHER OUTCOMES:
Genetic variant data | Up to 2 years
  Exploratory statistical genetic and bioinformatics analyses will be made using the data derived from the genomic sequencing to catalogue additional important variants and determine whether there are any patterns or associations among patient level risk factors, their outcomes and genomic information that was not identified by the original genomic sequencing analyses

CONTACTS AND LOCATIONS:
Overall Officials: Angela Alistar, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States